CLINICAL TRIAL: NCT02666521
Title: Study to Determine the Frequency and Associated Predictors of Hypoglycaemia in People With Type 2 Diabetes Mellitus Managed in Primary Care
Brief Title: Hypoglycaemia in People With Type 2 Diabetes in Primary Care
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: Primary Care Diabetes Society, UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0204; UKCRN ID 12188 (Other: UK Clinical Research Network)
Record Dates: First submitted 2016-01-20; First posted 2016-01-28 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2016-01

CONDITIONS: Diabetes Mellitus, Type 2; Hypoglycemia
Keywords: Primary Health Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite type 2 diabetes comprising the majority of cases of diabetes, the overall frequency of hypoglycaemia in this group has not been as carefully documented as in type 1 diabetes, particularly in relation to the clinical use of individual therapies in primary care.

The aim of this study is to provide robust data on the frequency and severity of hypoglycaemia in people with type 2 diabetes managed in primary care, and assess and explore associated risk factors.

DETAILED DESCRIPTION:
Background - previous studies have provided robust evidence on the link between intensive therapy and increased frequency of hypoglycaemia in people with type 1 diabetes. Despite type 2 diabetes comprising the majority of cases of diabetes, the overall frequency of hypoglycaemia in this group has not been as carefully documented as in type 1 diabetes, particularly in relation to the clinical use of individual therapies in primary care.

Recent prospective studies suggest that hypoglycaemia occurs more frequently than was previously thought for people with type 2 diabetes, particularly those treated with insulin and sulphonylureas. An increasingly elderly population, and earlier initiation of insulin and other newer therapies and treatment combinations, may influence the risk and severity of hypoglycaemic episodes.

The overall aim is to undertake research that provides robust data on the frequency and severity of hypoglycaemia in people with type 2 diabetes managed in primary care, and assess and explore associated risk factors.

PROSPECTIVE STUDY Aims - to prospectively evaluate the self-reported frequency and severity of hypoglycaemia in people with type 2 diabetes managed in primary care (stratified by participant treatment regime); to investigate the associated clinical and demographic predictors of hypoglycaemia.

Methods - we will undertake a prospective, observational cohort study. Firstly, general practices will be approached to participate in the study, with an aim of recruiting around 20 practices throughout the UK. All recruited sites will receive relevant study training for the purposes of recruiting participants and collecting/recording research data. Participating general practices will then identify potentially eligible individuals on their practice register; individuals will be invited via a study invitation pack sent in the post or given in person when they attend the practice. Individuals expressing an interest will be invited to attend an appointment at their general practice where informed consent will be obtained and baseline data collected (demographic, bio-medical and self-completion questionnaires). Participants will be provided with relevant study materials (glucose monitoring diaries, hypoglycaemia recording forms, and a blood glucose meter and strips) and asked to measure their blood glucose and record any episodes of hypoglycaemia, over a period of 12-months. Repeat biomedical and self-completion questionnaire data will be collected at 12-months follow-up.

The overall sample size for the prospective study is 422, based on recruiting a quota of participants on the following treatment regimens: 1) metformin only (n=62); 2) sulphonylurea based (n=140); 3) insulin based (n=140); and 4) incretin based (Dipeptidyl peptidase-4 (DPP4) or Glucagon-like peptide-1 (GLP-1)), (n=80). Practices will be asked to continue recruitment until targets are met for each of the treatment groups.

CROSS SECTIONAL STUDY Aim - to provide data on the prevalence of hypoglycaemia in people with type 2 diabetes who are managed in primary care and explore associated risk factors.

Methods - approach for participation will be made when potential volunteers attend for a planned appointment for diabetes care (e.g. diabetes annual review, diabetic retinopathy screening), through poster advertisement at the site. Their healthcare professional will also explain that there is a researcher at the clinic who is recruiting individuals with type 2 diabetes to take part in a research study. The researcher will then approach potential volunteers to provide a brief verbal explanation of the study, followed by a written participant information sheet for them to read. Subsequently, for individuals who volunteer to participate, they will be asked to sign a consent form and then given a questionnaire to self-complete (at their appointment or take home and post back to the research team). In addition, a researcher will obtain biomedical data from participants' medical records; no data will be collected until at least 48 hours has passed from the time informed consent was obtained, to allow time for participants who may change their mind about taking part.

The anticipated recruitment target for the cross-sectional study is to recruit up to 2000 participants.

ELIGIBILITY:
PROSPECTIVE STUDY

Inclusion Criteria:

* Confirmed diagnosis of type 2 diabetes mellitus
* Diagnosis at least 6 months prior to recruitment
* Registered at participating general practice
* Aged ≥ 18 years old
* On one of the following treatment regimens:

  1. metformin only
  2. sulphonylurea based (not on insulin or incretin-based therapy)
  3. insulin based (not on sulphonylurea, GLP-1 or DPP-4)
  4. incretin or incretin based therapy, DPP-4 or GLP-1 (not on sulphonylureas or insulin)
* HbA1c <9.0% at last reading Willingness to self-report episodes of hypoglycaemia and undertake home blood glucose self-monitoring for 12-months

Exclusion Criteria:

* Participant managed exclusively in secondary care
* Severe diabetic complications e.g. corrected visual acuity less than 6/12 in both eyes, major limb amputation or severe peripheral sensory neuropathy
* History of seizures unrelated to hypoglycaemia
* Severe systemic disease unrelated to diabetes
* Pregnancy
* Any reason why the participant may not be able to understand instructions or be unable or unwilling to co-operate with the study staff e.g. mental incapacity, language barriers

CROSS-SECTIONAL STUDY

Inclusion criteria:

* Confirmed diagnosis of type 2 diabetes mellitus
* Diagnosis at least 6 months prior to recruitment
* Registered at a general practice within Leicestershire, Rutland or Northamptonshire
* Treatment for type 2 diabetes includes oral hypoglycaemic drugs and/ or insulin

Exclusion criteria:

* Any reason why the participant may not be able to understand instructions or be unable or unwilling to co-operate with the study staff e.g. mental incapacity, language barriers
* Aged ≥ 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Type 2 diabetes managed in primary care
Sampling Method: Non-Probability Sample
Enrollment: 2327 (Actual)
Dates: Start 2012-07-20 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Frequency of mild hypoglycaemic episodes, compared by treatment regimen | at 12-months (Prospective)
  self-report
Frequency of mild hypoglycaemic episodes | Baseline (Cross-sectional);
  self-report

SECONDARY OUTCOMES:
Frequency of severe hypoglycaemic episodes, compared by treatment regimen | at 12-months (Prospective)
  self-report
Frequency of severe hypoglycaemic episodes | Baseline (Cross-sectional);
  self-report

OTHER OUTCOMES:
Hypoglycaemia symptoms | Baseline (Cross-sectional); Baseline and 12-months (Prospective)
  The Edinburgh Hypoglycaemia Scale
Awareness of hypoglycaemia | Baseline (Cross-sectional); Baseline and 12-months (Prospective)
  Hypoglycaemia Awareness Scale
Fear of hypoglycaemia | Baseline (Cross-sectional); Baseline and 12-months (Prospective)
  Hypoglycaemia Fear Survey
Health related quality of life | Baseline (Cross-sectional); Baseline and 12-months (Prospective)
  EQ-5D
Anxiety and depression | Baseline (Cross-sectional); Baseline and 12-months (Prospective)
  Hospital Anxiety and Depression Scale
Incidence and severity of hypoglycaemic episodes | up to 12-months (Prospective study group only)
  Hypoglycaemia recording form and diary

CONTACTS AND LOCATIONS:
Overall Officials: Prof Kamlesh Khunti, PhD, FRCGP, Principal Investigator — University of Leicester
Locations (1):
- Diabetes Research Centre, University of Leicester, Leicester, United Kingdom